CLINICAL TRIAL: NCT07239336
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate The Efficacy and Safety of DONQ52 in Active Celiac Disease Patients Who Have Duodenal Mucosal Damage and Persistent Symptoms Despite Attempting A Gluten-free Diet (DAISY STUDY)
Brief Title: Study of DONQ52 in Active Celiac Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DQB104CT
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + SIGE Gluten capsule (Placebo Comparator): Placebo subcutaneous (SC) injection as per protocol + SIGE Gluten capsule orally
  Interventions: Drug: Placebo DONQ52; Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) capsule
- DONQ52 + SIGE Gluten capsule (Experimental): DONQ52 subcutaneous (SC) injection as per protocol + SIGE Gluten capsule orally
  Interventions: Drug: DONQ52; Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) capsule

INTERVENTIONS:
Drug: Placebo DONQ52 — Placebo DONQ52 subcutaneous injection
  Arms: Placebo + SIGE Gluten capsule
Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) capsule — SIGE gluten capsules orally
  Arms: Placebo + SIGE Gluten capsule
Drug: DONQ52 — DONQ52 subcutaneous injection
  Arms: DONQ52 + SIGE Gluten capsule
Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) capsule — SIGE gluten capsules orally
  Arms: DONQ52 + SIGE Gluten capsule

SUMMARY:
The main aim is to see how DONQ52 works to improve small intestinal damage and reduce celiac-related symptoms due to gluten exposure, in participants with celiac disease (CeD) attempting to maintain a gluten-free diet (GFD) in treated participants versus placebo controls.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18 to 40 (kg/m2) at screening.
* Willingness to ingest a gluten-free product and Simulated Inadvertent Gluten Exposure (SIGE) products as per the study protocol.
* History of medically diagnosed, and adequately documented (i.e., included in the participant's medical records), CeD
* Attempting a GFD for at least 12 months prior to the screening visit.

  - The participants should be instructed not to alter dietary habits including a GFD during the study period.
* Valid results from central testing of blood documenting a positive result for the HLA DQ2.5 genotype (HLA-DQA1*05 and HLA-DQB1*02) (homozygous or heterozygous).
* Experienced at least 2 gluten-related symptom events (i.e., 2 different gluten-related symptoms which are diarrhea, abdominal pain, bloating, nausea, tiredness or 1 gluten-related symptom occurred twice) within a month before the screening.
* Willingness to undergo 2 on-study upper gastrointestinal endoscopies with duodenal biopsies.
* Presence of ongoing duodenal mucosal damage defined as Vh:Cd of 2.5 or less

Exclusion Criteria:

* Participants with documented history (i.e., included in the participant's medical records) of medically diagnosed Refractory Celiac Disease (RCD) or suspected RCD by the investigator.
* History of IgE-mediated reactions to wheat, barley, rye, or other ingredients in gluten-free and SIGE products used in this study (i.e., methylcellulose, and gelatin).
* History of cancer, including hematological malignancy and solid tumors, within 5 years prior to the screening visit, or history of T cell lymphoma or B cell lymphoma ever.
* History of hypersensitivity reactions including anaphylaxis to a biological medical product or any of the excipients.
* Participants who carry the HLA-DQ8 (HLA-DQA1*03 and DQB1*0302) genotype (homozygous or heterozygous).
* Any other chronic, active gastrointestinal disease (e.g., inflammatory bowel disease, microscopic colitis, eosinophilic esophagitis, peptic ulcer, gastroesophageal reflux disease, functional dyspepsia, or irritable bowel syndrome) that might in the investigator's opinion, interfere with the assessment of GI symptoms or small intestinal histology.
* Helicobacter pylori tests that indicate current infection.
* Positive either human immunodeficiency virus (HIV) antigen or antibody test at screening.
* Positive hepatitis B surface antigen (HBsAg) test or total hepatitis B core (HBc) antibody test at screening.
* Positive hepatitis C virus (HCV) antibody test at screening, except in participants who have negative results for HCV ribonucleic acid (RNA) test at screening.
* Positive for QuantiFERON-TB Gold test at screening that indicates active tuberculosis (TB) at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Villous Height to Crypt Depth Ratio (Vh:Cd) | Baseline to Week 27
  The Vh:Cd ratio represents mucosal architectural changes and a lower Vh:Cd ratio indicates more severe intestinal injury characterized by a flattening of the mucosa. The difference in the adjusted mean change from baseline (Run-in) to Week 27 in Vh:Cd between DONQ52 and placebo groups will be estimated using the analysis of covariance (ANCOVA) method. A negative change from baseline indicates worsening disease.

SECONDARY OUTCOMES:
Change in Average of total score of Celiac Disease Symptom Diary (CDSD) Gastrointestinal (GI) domain (abdominal pain, diarrhea, nausea, and bloating) calculated as two-week average. | Baseline to Week 27
  CDSD symptom severity score is an average of the daily symptom severity scores during the week. The daily symptom severity score is the average of the severity score for diarrhea, abdominal pain, bloating, nausea, and tiredness ranging from 0 to 4. Symptom severity is evaluated using 5-point Likert-type scales (none, mild, moderate, severe, and very severe). Higher scores indicate more severe symptoms. Results are reported as mean change from baseline at Week 13-14 and Week 25-26. A negative change from baseline indicates improvement.
Change in Average of the total score of non-stool GI symptoms (abdominal pain, nausea, and bloating) calculated as two-week average. | Baseline to Week 27
  CDSD GI symptom severity score is an average of the daily non-stool GI symptom severity scores during the week. The daily non-stool GI symptom severity score is the average of the severity score for abdominal pain, nausea, and bloating, ranging from 0 to 4. Symptom severity is evaluated using 5-point Likert-type scales (none, mild, moderate, severe, and very severe). Higher scores indicate more severe symptoms. Results are reported as mean change from baseline at Week 13-14 and Week 25-26. A negative change from baseline indicates improvement.
Change in Average of diarrhea frequency score as assessed by CDSD frequency supplement calculated as two-week average. | Baseline to Week 27
  Diarrhea frequency score assessed by CDSD frequency supplement is an average of the daily diarrhea frequency score during the week. Results are reported as mean change from baseline at Week 13-14 and Week 25-26. A negative change from baseline indicates improvement.
Relationship between the total score of CDSD GI domain and Patient Global Impression of Severity (PGI-S) or Patient Global Impression of Change (PGI-C). | Baseline to 47 weeks
  The PGI-S is a Patient-Reported Outcome (PRO) measure assessing participant's impression of overall severity of disease symptoms. The PGI-S consists of single-item which asks participant's disease severity over the past 7 days and 14 days. It is rated on a 5-point scale from None to Very Severe. This PGI-S has been specifically modified to focus on celiac disease symptoms (i.e., abdominal pain, bloating, diarrhea, and nausea), adapting the standard PGI-S framework to be celiac disease-specific.
  The PGI-C is a PRO measure assessing participant's impression of the overall change in disease symptoms. The PGI-C consists of single-item which asks the change of participant's clinical status since the start of the study. It is rated on a 7-point scale from Very Much Improved to Very Much Worse. This PGI-C has been specifically modified to focus on celiac disease symptoms (i.e., CDSD GI items), adapting the standard PGI-C framework to be celiac disease-specific.
Incidence and severity of adverse events (AEs) and their causal relationship to the investigational medicinal products (IMPs). | Baseline to 47 weeks
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a markedly abnormal physical examination finding, vital sign value, laboratory test value), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug.The investigator clinically judges whether an AE was caused by the IMP. This assessment of causality, often categorized as "related" or "not related," is a distinct step performed after an event has been identified and recorded as an AE.
Serum DONQ52 concentration. | Day1 to 47 weeks
Prevalence of anti-drug antibodies (ADAs) to DONQ52. | Day1 to 47 weeks
Incidence of anti-drug antibodies (ADAs) to DONQ52. | Day1 to 47 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chugai Pharmaceutical Co., Ltd., Study Director — clinical-trials@chugai-pharm.co.jp
Locations (3):
- United States (3):
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Novum Clinical Research, Clermont, Florida
  - Guardian Angel Research Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).